CLINICAL TRIAL: NCT00787124
Title: Transfusions and Nitric Oxide Level in Preterm Infants
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Children's Miracle Network (Other)
Responsible Party: Principal Investigator, Phillip Brian Smith, Associate Professor, Duke University
Other Study IDs: Pro00007939
Record Dates: First submitted 2008-11-06; First posted 2008-11-07 (Estimated); Results first posted 2014-01-15 (Estimated); Last update posted 2018-09-28 (Actual); Status verified 2018-08

CONDITIONS: Prematurity; Anemia; Necrotizing Enterocolitis
MeSH Terms: conditions — Premature Birth; Anemia; Enterocolitis, Necrotizing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood specimens for measurement of SNO-Hb. Samples will be discarded after measurement.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: < 28 weeks gestation, < 30 days of age, < 3 previous transfusions
- 2: < 28 weeks gestation, >=30 days of age, >= 3 previous transfusions

SUMMARY:
The purpose of this study is to better understand S-nitrosohemeglobin (SNO-Hb) in transfused blood of extremely preterm infants. The long term goal of the project is to identify variation in the SNO-Hb between packed red blood cell units, and between and among individual preterm infants pre and post-transfusion. Duke investigators are developing methods to replenish SNO-Hb, which, if successful, would improve RBC deformation in addition to providing a vasodilatory stimulation to hypoxic tissue, and lead to a randomized clinical trial testing treated vs. untreated RBC transfusions in extremely premature infants.

AIM 1. Measure the Total Hemoglobin (Hb)-bound nitric oxide (NO), Hb [Fe] NO, SNO-Hb (a calculated value = (total Hb-NO - Hb [Fe] NO) in blood to be transfused in extremely preterm babies, and in samples pre and post- transfusion from the babies.

Hypothesis 1: Measures of NO and SNO-Hb will be low in blood used for transfusion in preterm infants and will be decreased in the post-transfusion samples from the infants compared with the pre-transfusion samples.

AIM 2. Collect clinical data about study participants, including oxygen saturation and measures of perfusion pre and post-transfusion.

Hypothesis 2: Measures of perfusion will be reduced by 20% post-transfusion in extremely preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* Infant < 28 weeks gestation at birth
* Undergoing PRBC transfusion with a volume ≥ 10 cc/kg
* Availability and willingness of the parent/legally authorized representative to provide written informed consent.

Exclusion Criteria:

* Any concomitant condition, which in the opinion of the investigator would preclude a patient's participation in the study
* Previous participation in the study.

Max Age: 365 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants < 28 weeks gestation at birth undergoing a packed red blood cell transfusion
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2008-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: P Brian Smith, MD MHS, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- <30 Days: < 28 weeks gestation, < 30 days of age, < 3 previous transfusions
- >=30: < 28 weeks gestation, >=30 days of age, >= 3 previous transfusions
Period: Overall Study
Arm/Group | <30 Days | >=30
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | <30 Days | >=30 | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 4 | 8
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: days] | 20 (45) | 60 (37) | 40 (40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Secondary Outcome: Oxygen Saturation and Measures of Perfusion Pre and Post-transfusion.
Description: data not appropriately collected for the analysis due to machine malfunctions.
Time Frame: prior to, during, after transfusion
Arm/Group | <30 Days | >=30
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: SNOHgB Levels
Description: levels were never run by the laboratory
Time Frame: beginning and end of study
Arm/Group | <30 Days | >=30
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | <30 Days | >=30
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

LIMITATIONS AND CAVEATS:
no AE observed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No